CLINICAL TRIAL: NCT01239485
Title: Phase I Study of IRNEA (Irinotecan, Etoposide, Cytarabine) for Refractory or Relapsed Acute Leukemia in Children and Adolescents
Brief Title: Study of IRNEA (Irinotecan, Etoposide, Cytarabine) for Refractory or Relapsed Acute Leukemia in Children and Adolescents
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Korea Childhood Leukemia Foundation, Korea Childhood Leukemia Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLSG-0901, SNUCH-RAL-0901
Record Dates: First submitted 2010-11-08; First posted 2010-11-11 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Acute Leukemia
Keywords: Pediatric refractory or relapsed acute leukemia
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan (Experimental)
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — Chemotherapy: irinotecan, etoposide, and cytarabine daily for 5 days (on days 0, 1, 2, 3, & 4) -30 min: Atropin ivs 0 hour: irinotecan X mg/m2 in D5W 100 mL IV over 60 min 0 hour: etoposide 100 mg/m2 in x3 N/S mL IV over 60 min 12 hour: cytarabine 2,000 mg/m2 over 3 hr
  *if age ≤ 3 yrs: calculate all drugs in kg base (30kg=1m2) Irinotecan dose is escalated by 25-30% in successive cohorts. The starting irinotecan dose (level 1) is 20 mg/m2/dose on days 0 to 4.

SUMMARY:
The purpose of this study is to determine the maximum tolerable dose of irinotecan in combination with etoposide, cytarabine for refractory or relapsed acute leukemia in pediatric patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALL or AML.
* Prior therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  * ALL patients must have had two or more prior therapeutic attempts defined as

    * Persistent (BM blast>5%) initial disease after two induction attempts, or
    * Persistent (BM blast>5%) after re-induction attempt for first relapse or
    * Relapse after one re-induction attempt (2nd relapse)
  * AML patients must have one or more prior therapeutic attempts defined as

    * Refractory (BM blast>20%) initial disease after one induction attempts, or
    * Persistent (BM blast>5%) initial disease after two induction attempts, or
    * Relapse after one induction attempt (1st relapse)
  * Relapse after stem cell transplant: Patients are eligible 12 weeks after allogeneic stem cell transplant as long as patients are not actively being treated for GvHD and have recovered from transplant-related toxicities. Patients are eligible 8 weeks from the day of stem cell infusion for myeloablative autologous stem cell transplant, if hematological and all other eligibility criteria are met.
* Age: ≤ 21 years.
* Performance status: ECOG 0-2.
* Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

  1. Heart: a shortening fraction ≥ 28%
  2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
  3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
* Patients must lack any active viral infections or active fungal infection.
* Patients (or one of parents if patients age < 19) should sign informed

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant (except acute leukemia) or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.
4. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerable dose of irinotecan in combination with etoposide, cytarabine for refractory or relapsed acute leukemia in pediatric patient. | 28 days

SECONDARY OUTCOMES:
To evaluate the incidence and severity of toxicity and treatment related mortality. 2. To evaluate the response rate. 3. To determine the pharmacokinetic profile of irinotecan in combination with etoposide, cytarabine in pediatric patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D, ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea